CLINICAL TRIAL: NCT05315804
Title: Treatment of Intraosseous Periodontal Pockets by Non-surgical Therapy With Micro-instruments and Application of Amelogenins. A Randomized-controlled Clinical Trial
Brief Title: Treatment of Intraosseous Periodontal Defects With Amelogenins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Clinical Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 477/21
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Bone Loss; Periodontal Pocket
Keywords: Amelogenin; Periodontal Therapy; Periodontal Bone Loss; Intraosseous Bone Defect
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Pocket | interventions — Amelogenin

STUDY DESIGN:
Intervention Model Description: The study will be designed as a double-arm randomized controlled clinical trial. The intraosseous defects of subjects allocated in A group will be treated with MINSD and application of amelogenins in gel, while in B Group only MINSD will be performed. The null hypothesis of no statistically significant differences between the two modalities for the treatment of intraosseous defects will be tested.
Who Masked: Participant
Masking Description: Only patients will be unaware of the type of treatment performed, with prior written informed consent. So, they will be divided in the two groups of study after a process of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amelogenin Group (A) (Experimental): Amelogenins in gel will be applied in intraosseous periodontal defects, after Minimally Invasive Non Surgical Debridement (MINSD)
  Interventions: Other: MINSD and amelogenins
- No-amelogenin Group (B) (Active Comparator): Only Minimally Invasive Non Surgical Debridement (MINSD) will be performed
  Interventions: Other: MINSD

INTERVENTIONS:
Other: MINSD and amelogenins — After local anesthesia, MINSD will be performed using an ultrasonic scaler with fine tips and micro-curette; then, amelogenins in gel will be applied to the intraosseous periodontal pockets using a sterile syringe with plasticized needle.
  Arms: Amelogenin Group (A)
Other: MINSD — Only subgingival mechanical debridement (MINSD) will be performed with an ultrasonic scaler with fine tips and micro-curette.
  Arms: No-amelogenin Group (B)

SUMMARY:
The aim of the present investigation will be evaluate the healing of periodontal intraosseous defects following Minimally Invasive Non Surgical Debridement (MINSD) and application of amelogenins, compared to MINSD alone.

A total of 22 patients will be enrolled, selected by inclusion and exclusion criteria and randomly divided in two groups: amelogenin (A) and no-amelogenin group (B).

DETAILED DESCRIPTION:
The objective of the study will be compare the healing of periodontal intraosseous defects following treatment with Minimally Invasive Non Surgical Debridement (MINSD) and application of amelogenins compared to MINSD alone.

Twenty-two patients with intraosseous periodontal defects will be randomly assigned to treatment with MINSD and application of amelogenins (A Group) or MINSD alone (B Group).

Primary outcome will be "Clinical Attachment Level" (CAL) gain, while the secondary outcomes will be "Probing Depth" (PD), "Gingival Recession" (GR) and "Radiographic Defect Angle" (RDA).

After local anesthesia, in A group MINSD will be performed using an ultrasonic scaler with fine tips and micro-curette; then, amelogenins in gel will be applied in the intraosseous periodontal pockets using a sterile syringe with plasticized needle.

In the B group, only subgingival mechanical debridement (MINSD) will be performed with an ultrasonic scaler with fine tips and micro-curette.

Finally, a polishing paste will be applied to the supra-gingival level in both groups using a rubber cup. Patients of both groups will be recalled every month for professional oral hygiene and, after 6 months, all measurements will be repeated and the final evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis;
* Age ≥ 18 years old;
* Presence of at least 10 teeth per arch;
* Presence of at least two teeth with Probing Depth (PD) ≥ 5 mm per quadrant;
* Presence of at least one intraosseous pocket;
* Single-rooted and multi-rooted teeth.

Exclusion Criteria:

* Patients with systemic diseases;
* Prolonged antibiotic or anti-inflammatory treatment within 4 weeks prior to periodontal therapy;
* Pregnant or lactating;
* Tobacco smokers (≥ 10 cigarettes per day);
* Multi-rooted teeth with furcation involvement;
* Third molars.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of Clinical Attachment Level (CAL) gain (millimeters) | baseline and 6 months after periodontal therapy
  Distance from the cementoenamel junction to the bottom of the pocket

SECONDARY OUTCOMES:
Change of Probing Depth (PD) (millimeters) | baseline and 6 months after periodontal therapy
  Distance from the gingival margin to the bottom of the pocket
Change of Gingival Recession (GR) (millimeters) | baseline and 6 months after periodontal therapy
  Distance from gingival margin to the cementoenamel junction
Change of Radiographic Defect Angle (RDA) (grade °) | baseline and 6 months after periodontal therapy
  Radiographic intraosseous angle

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ramaglia, Principal Investigator — Federico II University
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No